CLINICAL TRIAL: NCT02994849
Title: OPTI-Prem: Optimising Neonatal Service Provision for Preterm Babies Born Between 27 and 31 Weeks of Gestation in England Using National Data, Qualitative Research and Economic Analysis
Brief Title: OPTI-Prem: Optimising Neonatal Service Provision for Preterm Babies Born Between 27 and 31 Weeks of Gestation in England
Acronym: OPTI-Prem
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: University of Leicester (Other); University of Oxford (Other); Neonatal Data Analysis Unit (Unknown); Imperial College London (Other); Bliss Charity (Other)
Responsible Party: Sponsor
Other Study IDs: 2016NEO87
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Neonatal Diseases and Abnormalities
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Premature babies, born several weeks before their due date, are often very ill in the first weeks and months of life, compared with those born at full term. Because babies' brains and bodies are still developing at this time, early birth puts them at increased risk of later problems with health and development. It is important to do everything possible to try to improve the overall health of these children. Not only will this help children and families, but it will also help to understand the correct amount and type of care they will need from the NHS in the future. At present, England has three types of neonatal units: Neonatal Intensive care units (NICUs) that can care for the most sick and most premature babies, Local Neonatal Units (LNUs) that generally care for slightly less sick babies, and Special Care baby units (SCBU) that care for larger premature babies who are generally well, but need time to grow and develop before going home.

For those premature babies born between 27 and 31 weeks of pregnancy, there is no information on whether they benefit from being looked after in one type of unit or another. At present there is no guidance, so these babies may be looked after in either LNUs or NICUs. Babies who are born at this stage of pregnancy cannot be looked after in a SCBU and sometimes need to be moved after birth to either a NICU or LNU. There are 84 LNUs and 45 NICUs in England. In 2014, about half of these babies were cared for in a NICU and half in a LNU. There is the need to know whether babies born between 27 and 31 weeks are best cared for in a NICU or LNU or if it does not matter.

The main things that control where a baby is born are where the mother has her antenatal care, and where there is a cot available for the baby. A mother may have antenatal care in a hospital that has a NICU, LNU or SCBU. Because it is difficult to predict which mother is going to have her baby early, she cannot be directed, at the time of her choosing her hospital for antenatal care, where to go to for care. There is uncertainty before birth which baby is likely to require intensive care, but usually the less mature babies need more intensive care.

In this study to find out where it is best to care for babies born at 27-31 weeks of pregnancy, the study will look at which type of unit: a) leads to the best outcome for babies born at each week of pregnancy in this range; b) is most cost-effective for families and the NHS and c) best considers views and needs of parents and staff caring for babies.

DETAILED DESCRIPTION:
Mixed methods, longitudinal study; 5 work streams, supported by a Parent Advisory Panel:

Work stream 1:Clinical Outcomes Study Using routinely collected data from the National Neonatal Research Database (NNRD) for babies born at 27-31 weeks of gestation, admitted to neonatal units in England 01/01/14-31/12/17.Estimates of differences in mortality and specified morbidities between babies cared for in LNUs and NICUs will be obtained Data will be linked to Hospital Episode Statistics (morbidity) and ONS(mortality) up to 1 year of age for longer term outcomes.

Work stream 2:Types of clinical care provided Using NNRD, data from a unit questionnaire (01/01/017-31/12/2017), and review of guidelines from neonatal units, variation in clinical practice in 6 areas will be examined: medical/nurse staffing; policies/practice re respiratory support; infection control, feeding and developmental care, discharge and length of stay. Where appropriate, outcomes (mortality, chronic lung disease, central line sepsis, receipt of breastmilk on discharge and length of stay in hospital) by week of gestational age, will be analysed between units with similar practices.

Work stream 3:Economic analysis A cost-effectiveness study comparing costs and outcomes of LNU versus NICU will be conducted.

Work stream 4:Ethnographic study with a representative group of parents and clinicians Observations and interviews will be used to explore factors parents think should guide decision making about place of care and how it happens in practice; clinicians' perspectives/practices on decision making and place of care; impact on parents/families of these decisions and subsequent change in care location; and how parents can best be supported at this time. 40 cases from 2 networks [20 real-time, 20 retrospective] will be studied.

Workstream 5:

Once the results of the 4 work streams are analysed, and conclusions reached, a working group will be set up in collaboration with BAPM to develop recommendations to be made available for health service delivery planning.

ELIGIBILITY:
Inclusion Criteria:

* preterm babies born at 27-31 weeks

Exclusion Criteria:

-

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm babies born at 27-31 weeks
Sampling Method: Non-Probability Sample
Enrollment: 4364 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year of age

CONTACTS AND LOCATIONS:
Overall Officials: Tilly Pillay, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

REFERENCES:
- [Result] Ismail AQT, Boyle EM, Pillay T; OptiPrem Study Group. The impact of level of neonatal care provision on outcomes for preterm babies born between 27 and 31 weeks of gestation, or with a birth weight between 1000 and 1500 g: a review of the literature. BMJ Paediatr Open. 2020 Mar 17;4(1):e000583. doi: 10.1136/bmjpo-2019-000583. eCollection 2020. PMID 32232179
- [Result] Cupit C, Paton A, Boyle E, Pillay T, Armstrong N; OPTI-PREM Study Team. Managerial thinking in neonatal care: a qualitative study of place of care decision-making for preterm babies born at 27-31 weeks gestation in England. BMJ Open. 2022 Jun 27;12(6):e059428. doi: 10.1136/bmjopen-2021-059428. PMID 35760541
- [Result] Pillay T, Modi N, Rivero-Arias O, Manktelow B, Seaton SE, Armstrong N, Draper ES, Dawson K, Paton A, Ismail AQT, Yang M, Boyle EM. Optimising neonatal service provision for preterm babies born between 27 and 31 weeks gestation in England (OPTI-PREM), using national data, qualitative research and economic analysis: a study protocol. BMJ Open. 2019 Aug 22;9(8):e029421. doi: 10.1136/bmjopen-2019-029421. PMID 31444186
- [Result] Cupit C, Paton A, Boyle E, Pillay T, Anderson J, Armstrong N; OPTI-PREM team. Parenting through place-of-care disruptions: A qualitative study of parents' experiences of neonatal care. Health Expect. 2024 Feb;27(1):e13933. doi: 10.1111/hex.13933. PMID 39102689
- [Result] Yang M, Campbell H, Pillay T, Boyle EM, Modi N, Rivero-Arias O. Neonatal health care costs of very preterm babies in England: a retrospective analysis of a national birth cohort. BMJ Paediatr Open. 2023 May;7(1):e001818. doi: 10.1136/bmjpo-2022-001818. PMID 37130654
- [Derived] Pillay T, Rivero-Arias O, Armstrong N, Seaton SE, Yang M, Banda VL, Dawson K, Ismail AQ, Bountziouka V, Cupit C, Paton A, Manktelow BN, Draper ES, Modi N, Campbell HE, Boyle EM. Optimising neonatal services for very preterm births between 27+0 and 31+6 weeks gestation in England: the OPTI-PREM mixed-methods study. Health Soc Care Deliv Res. 2025 Apr;13(12):1-126. doi: 10.3310/JYWC6538. PMID 40232009
- [Derived] Pillay T, Seaton SE, Yang M, Bountziouka V, Banda V, Campbell H, Dawson K, Manktelow BN, Draper ES, Modi N, Boyle EM, Rivero-Arias O; OPTI-PREM study group; Contributing neonatal units and leads. Improving outcomes for very preterm babies in England: does place of birth matter? Findings from OPTI-PREM, a national cohort study. Arch Dis Child Fetal Neonatal Ed. 2025 Aug 19;110(5):444-451. doi: 10.1136/archdischild-2024-327474. PMID 39730195
- See also: Clinical outcomes for babies born between 27 - 31 weeks of gestation: Should they be regarded as a single cohort? — https://doi.org/10.1016/j.jnn.2022.04.003
- See also: Improving outcomes for very preterm babies in England: does place of birth matter? Findings from OPTI-PREM, a national cohort study — https://fn.bmj.com/content/early/2025/03/02/archdischild-2024-327474
- See also: Cost-Effectiveness of Intensive and Local Neonatal Care Units in England: A Real-World Evidence Analysis of a National Birth Cohort — https://doi.org/10.1016/j.jval.2024.10.417
- See also: Exploring variation in quality of care and clinical outcomes between neonatal units: a novel use for the UK National Neonatal Audit Programme (NNAP) — https://bmjopenquality.bmj.com/content/11/4/e002017